CLINICAL TRIAL: NCT06686745
Title: A Phase I, First-in-Human, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0508 Monotherapy and Combination Therapy in Adult Participants With Locally Advanced/Metastatic Solid Tumors
Brief Title: Study of SIM0508 Alone and in Combination in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0508-101
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SIM0508 mono dose escalation (Experimental): Every 28 days is one cycle. Multiple dose levels of SIM0508 will be explored in dose escalation, and determine the maximum tolerated dose.
  Interventions: Drug: SIM0508 Tablets
- SIM0508 combination dose escalation (Experimental): Every 28 days is one cycle.Multiple dose levels of SIM0508 and olaparib will be explored in dose escalation, and determine the maximum tolerated dose.
  Interventions: Drug: SIM0508 in combination with olaparib
- SIM0508 in combination with olaparib (Experimental): Every 28 days is one cycle.Patients will be administered a potential recommended dose of SIM0508 combination with olaparib established from SIM0508 combination dose escalation.
  Interventions: Drug: SIM0508 in combination with olaparib

INTERVENTIONS:
Drug: SIM0508 Tablets — Every 28 days is one cycle. Multiple dose levels of SIM0508 will be explored in dose escalation, and determine the maximum tolerated dose.
  Arms: SIM0508 mono dose escalation
Drug: SIM0508 in combination with olaparib — Every 28 days is one cycle.Multiple dose levels of SIM0508 and olaparib will be explored in dose escalation, and determine the maximum tolerated dose.
  Arms: SIM0508 combination dose escalation
Drug: SIM0508 in combination with olaparib — Every 28 days is one cycle.Patients will be administered a potential recommended dose of SIM0508 combination with olaparib established from SIM0508 combination dose escalation.
  Arms: SIM0508 in combination with olaparib

SUMMARY:
This is a multicenter, open-label, first-in-human study to evaluate the safety,efficacy, and PK/PD characteristics of SIM0508 as a single agent and in combination with olaparib in participants with locally advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signature of informed consent form.
2. Participants with histologically confirmed ovarian cancer, prostate cancer,breast cancer , or pancreatic cancer.
3. ECOG score of 0 or 1.
4. Expected survival ≥ 12 weeks.

Exclusion Criteria:

1. Active hepatitis B (HBsAg or HBcAb positive and HBV DNA≥1×104 copies/mL or≥2000 international unit [IU]/mL) or hepatitis C (HCV antibody positive and HCV RNA≥ULN) infection; participant with HBsAg positive or detective HBV-DNA at screening should receive antiviral treatment as per local practice during the study.
2. Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
3. Participants unable to swallow study drug and participants with gastrointestinal disorders likely to interfere with absorption of the study drug.
4. Toxicities from previous anticancer therapies have not resolved (e.g to ≤ Grade 1).
5. Pregnant or nursing (lactating) women; other women of childbearing potential, unless the blood pregnancy test within 7 days of first dose of study drug is negative, and participants agree to use highly effective contraceptive methods from signing of informed consent to 180 days after the last dose of SIM0508 or olaparib, whichever comes later.
6. Male partinipants with female partners of reproductive potential, unless they agree to use highly effective contraceptive methods from signing of informed consent to 180 days after the last dose of SIM0508 and 90 days after the last dose of olaparib, whichever comes later.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  Primary Endpoints

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Chongqing Cancer Hospital, Chongqing